CLINICAL TRIAL: NCT07047040
Title: Analgesic Efficacy of Pre-operative Dose of Ketorolac And Gabapentin in Patients Undergoing Unilateral Total Knee Arthroplasty A Randomized Double Blinded Controlled Trial
Brief Title: Analgesic Efficacy of Pre-operative Dose of Ketorolac and Gabapentin
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour Shaaban Abdel-Aleem Mohamed, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pre-operative analgesia
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pain, Postoperative; Osteoarthritis, Knee
Keywords: total knee replacement; pre-operative analgesia; ketorolac; gabapentin
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — Ketorolac Tromethamine; Gabapentin

STUDY DESIGN:
Intervention Model Description: Patients scheduled for unilateral total knee replacement ranging from 40-80 years of age will be selected.
  Patients will be randomized into two groups. Experimental group will receive single dose of gabapentin 800 mg capsule and ketorolac 30 mg Ampule. While control group will receive normal saline ampule and empty capsule one hour prior to administration of spinal anesthesia.
  Pain will be assessed postoperatively by visual analogue score at,6 hours, 12 hours and 24 hours.
  total dose of analgesia in first 24 hours will be recorded. Any complications will be recorded in first 24 hours post- operative period.
  Follow up:
  Visual Analog Scale (VAS) will be used at 6, 12, 24 hours post-surgery for assessment of Pain. Any side effects or complications will be recorded. Time Up and Go (TUG) test after 24hrs post-operative. Oxford knee score (OKS) after 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Active Comparator): Experimental group will receive single dose of gabapentin 800 mg capsule and ketorolac 30 mg Ampule, one hour prior to administration of spinal anesthesia
  Interventions: Drug: Ketorolac Tromethamine 30 MG/ML Prefilled Syringe; Drug: Gabapentin
- control group (Placebo Comparator): control group will receive normal saline ampule and empty capsule one hour prior to administration of spinal anesthesia
  Interventions: Drug: Empty Medication Capsules

INTERVENTIONS:
Drug: Ketorolac Tromethamine 30 MG/ML Prefilled Syringe — a pre-operative dose of ketorolac and gabapentin is given to the patients undergoing unilateral TKA one hour prior to surgery, then a post-operative pain scores will be recorded
  Arms: Experimental group
Drug: Gabapentin — a pre-operative dose of ketorolac and gabapentin is given to the patients undergoing unilateral TKA one hour prior to surgery, then a post-operative pain scores will be recorded
  Arms: Experimental group
Drug: Empty Medication Capsules — two empty capsules of gabapentin
  Arms: control group

SUMMARY:
Evaluation of the analgesic efficacy of a pre-operative dose of ketorolac and gabapentin in reducing post-operative pain scores in patients undergoing TKA

DETAILED DESCRIPTION:
Elective total knee arthroplasty (TKA) is the gold standard for management of arthritis-associated pain and disability in osteoarthritis patients who have failed non-operative treatment modalitiesFollowing TKA, patients experience severe pain mediated by multiple pathways Painful stimuli to the body are detected by the free endings of peripheral nerves called nociceptors. Pre-emptive analgesia is analgesia given before the onset of painful stimuli to prevent central sensitization of nervous system to subsequent stimuli that could increase pain Studies have shown that pre-emptive analgesia reduce immediate postoperative pain and also prevent the development of chronic pain by decreasing altered sensory processing . Multimodal analgesia is the rational approach to pain management since no single analgesia targets all types of pain Multimodal analgesia, which is the use of at least 2 agents with differing mechanisms for pain control, has been shown to reduce hospital length of stay by 1.2 days and rehabilitation length of stay by 10 to 13 days compared with traditional postoperative analgesia. Ketorolac is a non-steroidal anti-inflammatory drug (NSAID). It is a cost-effective non selective cox inhibitor it inhibits prostaglandin biosynthesis. It is a potent analgesic with moderate anti-inflammatory.it inhibits platelet aggregation and increases bleeding time GABA analogues like Gabapentin is a structural analogue of gamma amino butyric acid, which was introduced in 1994 as an antiepileptic drug, particularly for partial seizures These drugs supress the hyper excitability of dorsal horn neurons caused due to tissue damage. They are also known to bind to the alpha 2 - delta subunit of voltage gated calcium channels and they have anxiolytic effect In this study we will assess the analgesic efficacy of pre-operative dose of combined ketorolac and Gabapentin in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients Undergoing Unilateral Total Knee Replacement from 40 years old to 80 years old

Exclusion Criteria:

* Rheumatoid Arthritis History of Renal impairment Patients refused to be enrolled in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluate the analgesic efficacy of a pre-operative dose of ketorolac and gabapentin in reducing post-operative pain scores in patients undergoing TKA. | during the first 24 hours post-operatively
  asses pain postoperatively at 6,12,24 hours using VAS score

SECONDARY OUTCOMES:
assess the impact of pre-operative ketorolac and gabapentin on post-operative opioid consumption | during the first 24 hours post-operatively
  by recording the total amount of opioids in both groups and comparing them
investigate the safety profile of pre-operative ketorolac and gabapentin | during the first 24 hours post-operatively
  by recording any side effects of these drugs during the study
evaluate the effect of pre-operative ketorolac and gabapentin on functional recovery | during the month after surgery
  by using Time UP and Go(TUG) Test in both groups and comparing them

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Mohamed Bakr, Professor, Study Director — Assiut University
Locations (1):
- Assiut University, Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skinner HB. Multimodal acute pain management. Am J Orthop (Belle Mead NJ). 2004 May;33(5 Suppl):5-9. PMID 15195936
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Hebl JR, Dilger JA, Byer DE, Kopp SL, Stevens SR, Pagnano MW, Hanssen AD, Horlocker TT. A pre-emptive multimodal pathway featuring peripheral nerve block improves perioperative outcomes after major orthopedic surgery. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):510-7. PMID 19258965
- [Background] Lee BH, Park JO, Suk KS, Kim TH, Lee HM, Park MS, Lee SH, Park S, Lee JY, Ko SK, Moon SH. Pre-emptive and multi-modal perioperative pain management may improve quality of life in patients undergoing spinal surgery. Pain Physician. 2013 May-Jun;16(3):E217-26. PMID 23703420